CLINICAL TRIAL: NCT06230133
Title: Feasibility and the Effects of Mindfulness-Based Stress Reduction (MBSR) on College Students' Resilience, Post-traumatic Stress Disorder Symptoms (PTSD) and Posttruamatic Growth (PTG)
Brief Title: Feasibility and the Effects of Mindfulness-Based Stress Reduction (MBSR) on College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Army Medical University, China (Other)
Responsible Party: Principal Investigator, Xiaofan Yan, lecturer, Army Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ArmyMedChina
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Posttraumatic Stress Symptom
Keywords: military medical students, mindfulness, resilience

STUDY DESIGN:
Intervention Model Description: Our study was designed as a controlled trial with a MBSR intervention and an control condition. Psychological data was assessed at baseline, at the end of the intervention, and one month later after the intervention, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness based stress reduction (MBSR) intervention (Experimental): MBSR intervention include 8 sessions. Each session took place once a week, 2 h per session, and lasted 8 consecutive weeks. Each session covered specific exercises and topics within the context of mindfulness practice and training. Participants were required to attend at least seven out of eight lessons, and to practice MBSR at least once per day as the homework. We provided participants with a series of audio recordings of MBSR exercises to help them do better. Participants were required to hand in the records of homework assignments before each intervention session, and they shared and discussed their homework assignments with other partners at the beginning of the intervention session. Additionally, the authors encouraged practitioners to develop an ability to bring mindfulness into the varied circumstances of daily living (e.g. Mindful running, mindful eating, mindful walking, and even mindful talking), especially stressful situations.
  Interventions: Behavioral: MBSR intervention
- Control condition (No Intervention): Participants in the control condition received university medical courses and physical training as usual.

INTERVENTIONS:
Behavioral: MBSR intervention — In our study, it is the same to arm description.
  Arms: mindfulness based stress reduction (MBSR) intervention

SUMMARY:
The goal of this retrospective control study is to learn about the effects of Mindfulness Based Stress Reduction (MBSR) intervention in military medical students' resilience, post-traumatic stress disorder symptoms (PTSD) and posttruamatic growth (PTG) etc. The main questions are aims to answer:

1. Would MBSR intervention improve psychological resilience, mindful attention awareness, satisfaction with life, and post-traumatic growth in military medical students？
2. Would MBSR intervention reduce anxiety, depression, and PTSD symptoms in military medical students？
3. Would the effects of MBSR intervention persist for at least one month in military medical students？ Participants in the intervention group will complete 8-week of MBSR training while those in the control group will not. Researchers will compare resilience, mindful attention awareness, satisfaction with life, and post-traumatic growth, etc. between the two groups.

DETAILED DESCRIPTION:
Recruitment for the study was done via broadcast email and posted notices online. 372 students filled out screening questionnaires and indicated their intention to participate the Mindfulness Based Stress Reduction (MBSR) course. We selected 120 students according to the participant criteria. Of the 120 participants, 60 were randomly assigned to the MBSR or control groups. However, 8 participants were absent more than two courses in the MBSR group, and 24 participants did not complete the post-test. Eventually, we enrolled 52 participants in the intervention group and 36 participants in the control group.

We designed a questionnaire survey on the internet to collect data. Two trained psychology teachers organized the survey at three time points: baseline (T0), the immediate postintervention (T1), and 1 month postintervention (T2).

Independent samples t-test and c2 analyses were used to test for possible group differences in demographic variables at baseline (T1).

Next, 2 (group) × 3 (time) mixed-model repeated-measure analysis of variance ( ANOVA) was conducted to determine the effect of MBSR. Effect sizes were reported as partial η² (ηp²) coefficients. To further interpret any time-by-group interactions, a series of t tests examined possible differences among baseline, post intervention and 1 month later after intervention.

ELIGIBILITY:
Inclusion Criteria:

* No regular meditation and yoga practice within the past 6 months;
* No current psychiatric symptoms and physical contraindications to exercise;
* the resilience scale scores were in the last 27% of the total 372 students.

Exclusion Criteria:

* Unwillingness to participant the mindfulness class;
* Absence from 2 or more classes;
* Do not complete the pre-, post-test and follow-up psychological assessment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The 10-item Connor-Davidson Resilience Scale (CD-RISC-10) | 12 weeks
  Item of CD-RISC-10 responses range from 0 ("not true at all") to 4 ("true nearly all of the time"). The overall score ranges from 0 to 40, with higher scores reflecting a greater ability to cope with adversity. The CD-RISC-10 showed excellent internal consistency in the current study, with Cronbach's alpha coefficients of 0.79, 0.87, and 0.92 at T0, T1, and T2, respectively.
The Posttraumatic Growth Inventory (PTG) | 12 weeks
  The Posttraumatic Growth Inventory (PTG) was developed to determine the positive changes that occur as a result of the traumatic events experienced by individuals. Participants were asked to rate the degree to which they experienced the change described by each item. The scale consists of 21 items in total and uses a 6-point Likert-type response scale ranging from 0 (almost never) to 5 (almost always). The total score ranged from 0 to 105, and the higher the score, the higher the level of PTG. Cronbach's Alpha for the total PTGI score was α = 0.95, 0.96, and 0.97 at T0, T1, and T2, respectively.
Satisfaction with Life Scale (SWLS) | 12 weeks
  In this study, life satisfaction was evaluated with the Satisfaction with Life Scale (SWLS). It consists of 5 items and each of them was rated on a 7-point Likert-type scale (1 = strongly disagree; 7 = strongly agree), and higher scores indicate higher life satisfaction. The Cronbach's α of the SWLS in this study was 0.84, 0.88, and 0.89 at T0, T1, and T2, respectively.
Mindful Attention Awareness Scale (MAAS) | 12 weeks
  Mindful Attention Awareness Scale (MAAS) is a self-reported questionnaire to assess dispositional mindfulness characterized by"open or receptive awareness of and attention" to the present moment. We used the Chinese version of the MAAS revised by Deng et al.. The MAAS included 15 items rated on a 6-point Likert scale ranging from 1 (almost always) to 6 (almost never). The total score ranged from 15 - 90, with higher scores indicating higher levels of mindfulness. The Cronbach's α of the MAAS in this study was 0.91, 0.91, and 0.95 at T0, T1, and T2, respectively.
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 12 weeks
  PTSD symptoms were assessed by the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) [33]. We adopted a revised Chinese version [34]in this study. 20 items assess the frequency and severity of PTSD symptoms regarding the index trauma, including symptom clusters of intrusion (Criterion B; 5 items), avoidance (Criterion C; 2 items), negative alterations of cognitions and mood (Criterion D; 7 items), and alterations in arousal and reactivity (Criterion E; 6 items). Participants indicated how much they have been bothered by each symptom using a 5-point scale from 0 (not at all) to 4 (extremely). Total scores range from 0 to 80, with a higher score indicating a greater level of posttraumatic stress. The total score ≥ 33 is considered positive. Cronbach's Alpha for the total PCL-5 in this study was 0.94, 0.93, and 0.96 at T0, T1, and T2, respectively.
Generalized Anxiety Disorder Scale (GAD-7) | 12 weeks
  Participants' anxiety was measured by the Generalized Anxiety Disorder Scale (GAD-7). It contains 7 items which drawn from the diagnostic criteria for GAD that had the strongest predictive validity with GAD as diagnosed by clinician interviews in a sample of 2740 patients across 15 clinics in the USA. Each item of GAD ranges from 0 (not at all) to 3 (nearly every day) and the total scores range from 0 to 21. A GAD-7 > 14 has been shown to have severe anxiety. Cronbach's Alpha for GAD-7 in this study was 0.89, 0.90, and 0.95 at T0, T1, and T2, respectively.
Patient Health Questionnaire (PHQ-9) | 12 weeks
  The Patient Health Questionnaire (PHQ-9) was used to assess depression severity. The scale contains 9 items. Response options for each item of the PHQ-9 score can range from 0 (not at all) to 3 (nearly every day). PHQ-9 total scores range from 0 to 27. A PHQ-9 score > 10 has been shown to have a sensitivity and specificity of 88% for major depression. Cronbach's Alpha for PHQ-9 in this study was 0.85, 0.87 and 0.89 at T0, T1, and T2, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Peng LI, professor, Study Director — Department of Military Psychology
Locations (1):
- Army Medical University, Chongqing, China